CLINICAL TRIAL: NCT00959881
Title: Combined Administration Of Begacestat And Donepezil: A Multiple-Dose Study In Healthy Subjects
Brief Title: Study Evaluating The Coadministration of Begacestat And Donepezil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 3183A1-1106; B1941005
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-04

CONDITIONS: Healthy Subjects
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil; begacestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil plus placebo (Experimental)
  Interventions: Drug: Donepezil plus placebo
- Donepezil plus begacestat (Experimental)
  Interventions: Drug: Donepezil; Drug: Begacestat

INTERVENTIONS:
Drug: Donepezil plus placebo — 5- and 10-mg tablets, single dose
  Other Names: Aricept
  Arms: Donepezil plus placebo
Drug: Donepezil — 5- and 10-mg tablets, single dose
  Other Names: Aricept
  Arms: Donepezil plus begacestat
Drug: Begacestat — 6 x 50-mg capsules, single dose
  Other Names: GSI-953, WAY-210953, PF-05212362
  Arms: Donepezil plus begacestat

SUMMARY:
This study examines the cardiac effects (effects on the heart) of administering donepezil and begacestat together to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Men and women of non-childbearing potential
* Non smoker or smoker of <10 cigarettes per day and able to refrain from smoking during study
* 18-50 years old

Exclusion Criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Cardiac rhythm abnormalities
* Family history of cardiac risk factors

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic interaction of multiple doses of begacestat and donepezil coadministered to healthy subjects as assessed by 12-lead electrocardiogram (ECG). | 5 months

SECONDARY OUTCOMES:
Pharmacokinetic parameters including Cmax, AUC, and t 1/2 | 5 months
Safety and tolerability as assessed by results of 12-lead ECGs, cardiac telemetry, laboratory tests, vital signs, physical examinations and reported adverse events. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3183A1-1106&StudyName=Study%20Evaluating%20The%20Coadministration%20of%20Begacestat%20And%20Donepezil